CLINICAL TRIAL: NCT03152552
Title: A Multi-center, Randomized, Double-blind, Parallel-group Dose-finding Study to Assess the Effect of 3 Doses of LIK066 Compared to Placebo or Empagliflozin in Type 2 Diabetes Mellitus Patients With Heart Failure
Brief Title: A Dose Finding Study to Assess the Effect of LIK066 Compared to Placebo or Empagliflozin in Patients With Type 2 Diabetes Mellitus and Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study terminated prematurely because of slow enrollment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIK066B2204; 2016-003084-19 (EudraCT Number)
Record Dates: First submitted 2017-05-08; First posted 2017-05-15 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus and Heart Failure
Keywords: Diabetes mellitus; LIK066; Obesity; Type 2 diabetes mellitus (T2DM); Heart Failure (HF); Hypertension; Renal dysfunction; Adult-onset diabetes; Noninsulin-dependent diabetes mellitus (NIDDM); High blood sugar
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure; Obesity; Diabetes Mellitus, Type 2; Hypertension; Renal Insufficiency; Hyperglycemia | interventions — licogliflozin; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LIK066 2.5mg (Experimental): Eligible participants randomized to this treatment arm received the LIK066 2.5mg dose regimen once daily for 36 weeks.
  Interventions: Drug: LIK066
- LIK066 10mg (Experimental): Eligible participants randomized to this treatment arm received the LIK066 10mg dose regimen once daily for 36 weeks.
  Interventions: Drug: LIK066
- LIK066 50mg (Experimental): Eligible participants randomized to this treatment arm received the LIK066 50mg dose regimen once daily for 36 weeks.
  Interventions: Drug: LIK066
- Empagliflozin (Active Comparator): Participants randomized to this treatment arm received empagliflozin once daily for 36 weeks.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Participants randomized to this treatment arm received LIK066 matching placebo and empagliflozin matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIK066 — LIK066 was supplied in different doses as tablets taken orally.
  Arms: LIK066 10mg; LIK066 2.5mg; LIK066 50mg
Drug: Placebo — Placebo was supplied as tablets and capsules taken orally.
  Arms: Placebo
Drug: Empagliflozin — Empagliflozin was supplied as capsules taken orally.
  Arms: Empagliflozin

SUMMARY:
This was a dose-finding study to evaluate the efficacy, safety and tolerability of 3 different doses of LIK066 compared to placebo or empagliflozin in T2DM patients with heart failure

DETAILED DESCRIPTION:
The study was prematurely discontinued on 04-May-2018 due to slow enrollment that would preclude obtaining study results in a timely manner.

ELIGIBILITY:
Key Inclusion Criteria:

* BMI ≥ 22kg/m^2
* Type 2 diabetes with HbA1c between 6.5% and 10.0%
* Documented symptomatic chronic heart failure (NYHA II-IV)
* Plasma NT-proBNP > 300pg/ml
* eGFR ≥ 45ml/min/1.73m^2 (calculated by MDRD)

Key Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Type 1 diabetes, monogenic diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes
* History of ketoacidosis, lactic acidosis, or hyperosmolar coma
* Symptomatic genital infection or UTI within 4 weeks of screening
* Myocardial infarction, stroke, surgery for heart disease, percutaneous coronary intervention within 3 months of randomization
* Unstable angina within 3 months of screening
* Isolated right HF due to pulmonary disease
* Patients with a mean sitting systolic blood pressure ≤ 100mmHg, at randomization
* History of lower limb amputation
* Diabetic foot ulcer at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (98):
- United States (21):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Carmichael, California
  - Novartis Investigative Site, Concord, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Delray Beach, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Gurnee, Illinois
  - Novartis Investigative Site, Bogalusa, Louisiana
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Sugar Land, Texas
  - Novartis Investigative Site, Tacoma, Washington
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
  - Novartis Investigative Site, Buenos Aires
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Lennik, Brussels Capital
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (6):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint-Jérôme, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Croatia (3):
  - Novartis Investigative Site, Krapinske Toplice
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Zagreb
- Czechia (7):
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Svitavy, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Fryštát
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Přerov
- Denmark (2):
  - Novartis Investigative Site, Hellerup
  - Novartis Investigative Site, Svendborg
- Germany (6):
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Stuttgart
- Hungary (4):
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szekszárd
- Ireland (3):
  - Novartis Investigative Site, Wilton, Cork
  - Novartis Investigative Site, County Limerick
  - Novartis Investigative Site, Dublin
- Italy (5):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, San Donato Milanese, MI
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Rimini
- Novartis Investigative Site, Durango, Mexico
- Netherlands (4):
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Utrecht
  - Novartis Investigative Site, Venlo
- Norway (3):
  - Novartis Investigative Site, Loerenskog
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Trondheim
- Poland (2):
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Ponce, Puerto Rico
- Novartis Investigative Site, Singapore, Singapore
- South Africa (3):
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Paarl, Western Cape
  - Novartis Investigative Site, Worcester
- South Korea (4):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Valencia, Valencia
- Taiwan (3):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- United Kingdom (4):
  - Novartis Investigative Site, Chelmsford, Essex
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, Sunderland, Tyne and Wear
  - Novartis Investigative Site, Birmingham

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized in a 1:1:2:2:2 ratio to one of 5 regimens (LIK066 2.5mg, 10mg, 50 mg, EMPA 25mg, Pbo) at Visit 201 (randomization) with a plan to be treated for 36 weeks.
Pre-assignment Details: A placebo run-in period (Epoch 2) running up to 2 weeks before randomization was used to assess eligibility
Groups:
- LIK066 2.5mg: LIK066 2.5mg once daily
- LIK066 10mg: LIk066 10mg once daily
- LIK066 50mg: LIK066 50mg once daily
- EMPA 25mg: Empagliflozin 25 mg once daily
- Placebo: LIK066 matching placebo and empagliflozin matching placebo
Period: Treatment Period 1 (12 Weeks)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Started (Randomized Set (RAN): all randomized patients) | 15 | 16 | 31 | 30 | 33
Full Analysis Set (FAS) (All patients in RAN who were not mis-randomized) | 15 | 16 | 30 | 30 | 33
Completed (Completed EPOCH 3 (double-blind period 1)) | 7 | 5 | 10 | 10 | 12
Not Completed | 8 | 11 | 21 | 20 | 21
Not completed — Death | 0 | 1 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 8 | 9 | 19 | 19 | 20
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Technical problems | 0 | 0 | 1 | 0 | 0
Not completed — Subject/guardian decision | 0 | 0 | 0 | 1 | 0
Period: Treatment Period 2 (24 Weeks)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Started | 7 | 5 | 9 (All patients who entered Treatment Period 2 (EPOCH 4)) | 9 (All patients who entered Treatment Period 2 (EPOCH 4)) | 11 (All patients who entered Treatment Period 2 (EPOCH 4))
Completed (Completed EPOCH 4 (double-blind period 2)) | 1 | 0 | 0 | 0 | 0
Not Completed | 6 | 5 | 9 | 9 | 11
Not completed — Study terminated by sponsor | 6 | 5 | 9 | 9 | 11

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics and efficacy analyses were done on Full Analysis Set (FAS). One patient from the LIK066 50 mg group, was misrandomized,and had not taken any study medication and thus was excluded from the Full analysis set (FAS) and the Safety analysis set (SAF).
Groups:
- Total: Total of all reporting groups
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 30 | 30 | 33 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (7.10) | 69.8 (9.69) | 65.8 (9.08) | 68.6 (7.89) | 67.8 (10.93) | 67.8 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 6 | 10 | 14 | 35
  Male | 14 | 12 | 24 | 20 | 19 | 89
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 14 | 14 | 28 | 28 | 29 | 113
  Black | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 2 | 2 | 1 | 3 | 9
  Other | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) at Week 12
Description: Evaluation of NT-proBNP was performed by a central laboratory. For Change from baseline, Geometric mean is the geometric mean of the endpoint to baseline ratio. Pre-planned statistical analysis was not performed for this primary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized. LIK066 doses and placebo arms are considered per study primary objective.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | Placebo
Number analyzed (Participants) | 9 | 8 | 12 | 16
ratio | 0.8 [0.5 to 1.2] | 0.6 [0.2 to 1.7] | 0.8 [0.7 to 1.1] | 1.1 [0.8 to 1.6]

2. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Weeks 12 and 36
Description: HbA1c was measured from a blood sample and analyzed using a National Glycohemoglobin Standardization Program (NGSP) certified method at a central laboratory. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 9 | 8 | 12 | 14 | 18
Percentage (%)
  Change from BL at Week 12 | -0.29 (0.836) | -0.01 (0.508) | -0.58 (0.335) | -0.44 (1.176) | -0.04 (0.913)
  Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 3
  Change from BL at Week 36 | 0.13 (0.961) |  | -0.60 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -1.83 (0.321)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 12 and 36
Description: FPG was measured from a blood sample after an overnight fast; patients were not allowed to eat or drink anything (except water) for at least 8 h before each study visit. Samples were analyzed at a central laboratory. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized.
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/L)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 8 | 6 | 12 | 13 | 15
millimoles per litre (mmol/L)
  Change from BL at Week 12 | -1.021 (1.0368) | -2.041 (4.9772) | -0.426 (2.1451) | -1.303 (2.4386) | -1.187 (3.9653)
  Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 3
  Change from BL at Week 36 | 0.392 (1.1119) |  | -1.200 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -4.733 (0.3055)

4. Secondary Outcome: Change From Baseline in Body Weight at Weeks 12 and 36
Description: Body weight was measured to the nearest 0.1 kg on a calibrated scale (weight and bio-impedance measurements), provided by the sponsor. Exceptionally (e.g. if the body weight exceeded the limits of the provided scale) sites were allowed to use another scale for weight measurement as available, but during the study the same scale was to be used for the same patient. The measurement was performed with the study patient in underwear and without shoes. Indoor clothing was also acceptable, but measurements were to be done consistently (either with underwear or with indoor clothing) throughout the study. Voiding before weight measurement was required. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 9 | 8 | 13 | 14 | 18
kilogram (kg)
  Change from BL at Week 12 | -0.78 (2.734) | -1.83 (1.402) | -2.15 (2.397) | -2.25 (1.894) | -0.34 (2.115)
  Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 3
  Change from BL at Week 36 | -2.21 (1.586) |  | -3.90 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 0.47 (6.158)

5. Secondary Outcome: Change From Baseline in Body Composition Assessed by Bio-impedance (Total Body Fat Mass) at Weeks 12 and 36
Description: Body composition was measured in all patients using bio-impedance, except in patients where it was contra-indicated, e.g. those using an implantable cardioverter-defibrillator. Body composition parameters were assessed as available for the different models of calibrated bio-impedance scales. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized.
Measure: Mean (Standard Deviation); unit: Percentage of body fat mass
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 6 | 7 | 11 | 12 | 15
Percentage of body fat mass
  Wk 12 Chge from BL | -0.77 (2.276) | -1.51 (5.048) | -0.32 (4.675) | 1.63 (3.639) | -1.77 (7.812)
  Wk 36 Chge from BL: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2
  Wk 36 Chge from BL | 2.25 (1.485) |  | 0.20 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 6.70 (20.082)

6. Secondary Outcome: Change From Baseline in Body Composition Assessed by Bio-impedance (Visceral Fat Level) at Weeks 12 and 36
Description: Body composition was measured in all patients using bio-impedance, except in patients where it was contra-indicated, e.g. those using an implantable cardioverter-defibrillator. Body composition parameters were assessed as available for the different models of calibrated bio-impedance scales. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented. Visceral fat levels were measured by Omron device. Levels ranged from 1 - 30 and are relative (not absolute) values. The Omron scale values are: 0 - 9 (normal), 10 - 14 (high) and 15 - 30 (very high). Visceral fat area ( 0 - approx. 300cm^2, 1 inch = 2.54 cm) distribution with 30 levels.
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized.
Measure: Mean (Standard Deviation); unit: Level
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 15
Level
  Wk 12 Chge from BL | -2.429 (4.6853) | -2.857 (3.8914) | -0.436 (4.6877) | -0.417 (1.3114) | -3.200 (4.7988)
  Wk 36 Chge from BL: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2
  Wk 36 Chge from BL | 0.000 (1.4142) |  | 0.000 (NA) — N/A: Not estimable due to insufficient number of participants with events |  | 3.500 (7.7782)

7. Secondary Outcome: Change From Baseline in Body Composition Assessed by Bio-impedance (Lean Body Mass) at Weeks 12 and 36
Description: as for outcome 5
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized.
Measure: Mean (Standard Deviation); unit: Percentage of body fat mass
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 6 | 6 | 10 | 12 | 14
Percentage of body fat mass
  Wk 12 Chge from BL | -2.32 (7.063) | -2.32 (5.774) | -0.24 (2.022) | -0.68 (2.454) | 1.64 (4.584)
  Wk 36 Chge from BL: number analyzed (Participants) | 2 | 0 | 1 | 0 | 2
  Wk 36 Chge from BL | -0.85 (1.344) |  | -0.30 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -5.35 (13.223)

8. Secondary Outcome: Change From Baseline in Body Composition Assessed by DXA (Total Body Fat Mass) at Weeks 12 and 36
Description: A whole body DXA scan was performed to assess Total Body Fat Mass (Whole Body Minus Head Hologic, Whole Body Minus Head Lunar). DXA data were transferred to a central reading vendor for independent review and analysis. Only descriptive statistics done.
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized. The analysis included patients who participated in the DXA sub-study. Due to early termination of the study, only the data shown was available.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 1 | 0 | 4 | 4 | 1
kilogram (kg)
  BL Whole Body Minus Head Hologic: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1
  BL Whole Body Minus Head Hologic | 35.970 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  | 18.870 (NA) — NA: Not estimable due to insufficient number of participants with events | 27.550 (NA) — NA: Not estimable due to insufficient number of participants with events
  Wk 12 Whole Body - Hd Hologic Chge BL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Wk 12 Whole Body - Hd Hologic Chge BL | -0.310 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |  | -4.280 (NA) — NA: Not estimable due to insufficient number of participants with events
  Wk 36 Whole Body - Hd Hologic Chge BL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Wk 36 Whole Body - Hd Hologic Chge BL | -3.800 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |  | -5.590 (NA) — NA: Not estimable due to insufficient number of participants with events
  BL Whole Body Minus Head Lunar: number analyzed (Participants) | 0 | 0 | 3 | 2 | 0
  BL Whole Body Minus Head Lunar |  |  | 29.350 (4.9403) | 37.455 (6.0175) |
  Wk 12 Whole Body - Hd Lunar Chge BL: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Wk 12 Whole Body - Hd Lunar Chge BL |  |  | -1.260 (NA) — NA: Not estimable due to insufficient number of participants with events | 1.190 (NA) — NA: Not estimable due to insufficient number of participants with events |
  Wk 36 Whole Body - Hd Lunar Chge BL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Body Composition Assessed by DXA (Visceral Fat Mass) at Weeks 12 and 36
Description: A whole body DXA scan was performed to assess Visceral Fat Mass (Whole Body Minus Head Hologic, Whole Body Minus Head Lunar). DXA data were transferred to a central reading vendor for independent review and analysis. Only descriptive statistics done.
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized. The analysis included patients who participated in the DXA sub-study. Due to early termination of the study, no data was collected.
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Body Composition Assessed by DXA (Lean Body Mass) at Weeks 12 and 36
Description: A whole body DXA scan was performed to assess Lean Body Mass (Whole Body Minus Head Hologic, Whole Body Minus Head Lunar). DXA data were transferred to a central reading vendor for independent review and analysis. Only descriptive statistics done.
Time Frame: Baseline, Week 12, Week 36
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 1 | 0 | 4 | 4 | 1
kilogram (kg)
  Wk 12 Whole Body - Hd Hologic Chge BL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Wk 12 Whole Body - Hd Hologic Chge BL | -1.910 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |  | 4.980 (NA) — NA: Not estimable due to insufficient number of participants with events
  Wk 36 Whole Body - Hd Hologic Chge BL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Wk 36 Whole Body - Hd Hologic Chge BL | 0.860 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |  | 1.700 (NA) — NA: Not estimable due to insufficient number of participants with events
  Wk 12 Whole Body - Hd Lunar Chge BL: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Wk 12 Whole Body - Hd Lunar Chge BL |  |  | -1.290 (NA) — NA: Not estimable due to insufficient number of participants with events | -2.960 (NA) — NA: Not estimable due to insufficient number of participants with events |
  Wk 36 Whole Body - Hd Lunar Chge BL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Body Composition Assessed by DXA (Total Body Water) at Weeks 12 and 36
Description: A whole body DXA scan was performed to assess Total Body Water (Whole Body Minus Head Hologic, Whole Body Minus Head Lunar). DXA data were transferred to a central reading vendor for independent review and analysis. Only descriptive statistics done.
Time Frame: Baseline, Week 12, Week 36
Population: FAS consisted of all randomized patients who were not mis-randomized. Analysis included patients who participated in the DXA sub-study. Due to early termination of the study, no data was collected.
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Weeks 12 and 36
Description: Three sitting BP measurements were performed. At each visit, sitting BP was derived as the mean of three readings of the sitting SBP/DBP at that visit. Pre-planned statistical analyses were not performed for these secondary endpoints due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized. Due to early termination of the study, only the data shown was available.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 9 | 8 | 13 | 14 | 18
millimeter of mercury (mmHg)
  SBP Change from BL at Week 12 | 5.15 (13.485) | 0.17 (15.373) | -9.54 (16.884) | -6.98 (15.031) | -2.85 (11.967)
  SBP Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 3
  SBP Change from BL at Week 36 | 13.78 (17.900) |  | -4.00 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 0.00 (8.627)
  DBP Change from BL at Week 12 | -2.00 (6.582) | 4.50 (12.746) | -4.46 (11.238) | -1.81 (10.421) | -2.00 (8.596)
  DBP Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 3
  DBP Change from BL at Week 36 | 1.12 (3.975) |  | 3.66 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -0.44 (8.517)

13. Secondary Outcome: Change From Baseline in Fasting Lipid Profile (Triglycerides (TG)) at Weeks 12 and 36
Description: TG was measured on blood samples obtained after an overnight fast and analyzed at a central laboratory. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 9 | 6 | 12 | 13 | 15
Percent change
  % Change from BL at Week 12 | -1.623 (35.2838) | 19.089 (31.4798) | 9.878 (30.3065) | 8.865 (35.0872) | -2.979 (25.1049)
  % Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 3
  % Change from BL at Week 36 | 4.324 (31.4438) |  | 14.286 (NA) — NA: Not estimable due to insufficient number of participants with events |  | -1.111 (18.3586)

14. Secondary Outcome: Change From Baseline in Fasting Lipid Profile (Lipoproteins) at Weeks 12 and 36
Description: Lipoproteins (High Density Lipoprotein (HDL) Cholesterol, Low Density Lipoprotein (LDL) Cholesterol) were measured on blood samples obtained after an overnight fast and analyzed at a central laboratory. Pre-planned statistical analysis were not performed for these secondary endpoints due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 9 | 8 | 7 | 12 | 12
Percent change
  HDL % Change from BL at Week 12 | 9.33 (16.735) | -10.54 (20.590) | 0.26 (9.772) | 2.18 (12.179) | -0.67 (13.322)
  HDL % Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 2
  HDL % Change from BL at Week 36 | 10.70 (16.257) |  | 0.00 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 35.00 (49.497)
  LDL % Change from BL at Week 12 | 22.02 (35.466) | 2.62 (17.525) | 16.40 (36.928) | 22.24 (35.145) | -1.59 (31.970)
  LDL % Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 2
  LDL % Change from BL at Week 36 | 22.73 (31.690) |  | -3.57 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 0.22 (13.163)

15. Secondary Outcome: Change From Baseline in Fasting Lipid Profile (Total Cholesterol) at Weeks 12 and 36
Description: Total Cholesterol was measured on blood samples obtained after an overnight fast and analyzed at a central laboratory. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: FAS consisted of all randomized patients who were not mis-randomized. Analysis included patients who participated in the study. Due to early termination of the study, only the data shown was available. 'Overall Number of Participants Analyzed' = enrolled in the study. 'Number Analyzed' = number of participants with data available.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 9 | 8 | 7 | 12 | 12
Percent change
  % Change from BL at Week 12 | 9.69 (23.892) | -2.66 (13.202) | 6.32 (22.667) | 10.83 (11.330) | 1.46 (16.741)
  % Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 2
  % Change from BL at Week 36 | 14.72 (13.147) |  | 2.04 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 10.27 (28.326)

16. Secondary Outcome: Change From Baseline in High Sensitive C-reactive Protein (hsCRP) at Weeks 12 and 36
Description: hs-CRP is an inflammation biomarker. For Change from baseline, Geometric mean is the geometric mean of the endpoint to baseline ratio. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: milligram per litre (mg/L)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 11 | 10
milligram per litre (mg/L)
  Change from BL at Week 12 | 0.543 [0.086 to 3.446] | 0.722 [0.157 to 3.321] | 1.997 [0.758 to 5.263] | 0.714 [0.353 to 1.443] | 1.018 [0.661 to 1.566]
  Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 0 | 3
  Change from BL at Week 36 | 0.953 [0.221 to 4.112] |  | 0.620 [NA to NA] — NA: Not estimable due to insufficient number of participants with events |  | 0.578 [0.172 to 1.945]

17. Secondary Outcome: Change From Baseline in 24 Hour Urinary Glucose Excretion (UGE) at Weeks 12 and 36
Description: UGE was measured from a 24h urine collection from about 25% of randomized patients and analyzed at a central laboratory. Only descriptive analysis done.
Time Frame: Baseline, Week 12, Week 36
Population: FAS consisted of all randomized patients who were not mis-randomized. Due to early termination of the study, only the data shown was available. 'Overall Number of Participants Analyzed' = enrolled in the 24 hour urine collection sub-study. 'Number Analyzed' = number of participants with data available.
Measure: Mean (Standard Deviation); unit: millimoles per 24 hours (mmol/24h)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 5
millimoles per 24 hours (mmol/24h)
  Change from BL at Week 12 | 256.245 (129.0682) | 346.360 (107.3671) | 305.110 (NA) — NA: Not estimable due to insufficient number of participants with events | 254.270 (198.8243) | 84.778 (222.6565)
  Change from BL at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in 24 Hour Sodium Excretion at Weeks 12 and 36
Description: Sodium excretion was measured from a 24h urine collection from about 25% of randomized patients and analyzed at a central laboratory. Only descriptive statistics were done.
Time Frame: Baseline, Week 12, Week 36
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: millimoles per 24 hours (mmol/24h)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7
millimoles per 24 hours (mmol/24h)
  Change from BL at Week 12 | -38.5 (86.69) | 45.6 (40.52) | -42.6 (28.50) | 82.3 (98.29) | -43.9 (112.48)
  Change from BL at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Change From Baseline in Left Atrial Size at Weeks 12 and 36
Description: A limited two-dimensional and Doppler ECHO examination was performed to assess ECHO parameters. The images were sent to a central reading vendor for independent review and analysis. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized. LIK066 doses and placebo arms were considered per study objective. Due to early termination of the study, only the data shown was available.
Measure: Mean (Standard Deviation); unit: milliliter per square meter (mL/m^2)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | Placebo
Number analyzed (Participants) | 3 | 4 | 7 | 11
milliliter per square meter (mL/m^2)
  Change from BL at Week 12 | -1.167 (14.8123) | 0.075 (6.7884) | 2.700 (7.2155) | -1.045 (11.0223)
  Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 3
  Change from BL at Week 36 | 16.333 (20.9194) |  | 0.300 (NA) — NA: Not estimable due to insufficient number of participants with events | 5.100 (6.2960)

20. Secondary Outcome: Change From Baseline in Left Atrial Volume at Weeks 12 and 36
Description: A limited two-dimensional and Doppler ECHO examination was performed to assess ECHO parameters. The images were sent to a central reading vendor for independent review and analysis.Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | Placebo
Number analyzed (Participants) | 5 | 4 | 8 | 11
milliliter (mL)
  Change from BL at Week 12 | 12.360 (42.7067) | 0.225 (15.4157) | 7.725 (16.9351) | -3.591 (22.8382)
  Change from BL at Week 36: number analyzed (Participants) | 3 | 0 | 1 | 3
  Change from BL at Week 36 | 34.800 (51.0409) |  | -0.900 (NA) — NA: Not estimable due to insufficient number of participants with events | 11.333 (12.7892)

21. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Class I, II, II or IV
Description: The NYHA Functional Classification classifies patients' heart failure according to the severity of their symptoms. The classification is as follows: Class I: no limitation of physical activity, ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath); Class II: slight limitation to physical activity, comfortable at rest, ordinary physical activity results in fatigue, palpitation or dyspnea; Class III: marked limitation of physical activity, comfortable at rest, less than ordinary activity causes fatigue, palpitation or dyspnea; Class IV: unable to carry on any physical activity without discomfort, symptoms of heart failure at rest, if any physical activity is undertaken, discomfort increases. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 12, Week 36
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | Placebo
Number analyzed (Participants) | 9 | 8 | 13 | 18
Participants
  Week 12: Class l | 1 | 1 | 1 | 1
  Week 12: Class ll | 6 | 6 | 10 | 13
  Week 12: Class lll | 2 | 1 | 2 | 4
  Week 12: Class lV | 0 | 0 | 0 | 0
  Week 36: number analyzed (Participants) | 3 | 0 | 1 | 3
  Week 36: Class l | 0 | 0 | 0 | 0
  Week 36: Class ll | 3 | 0 | 1 | 3
  Week 36: Class lll | 0 | 0 | 0 | 0
  Week 36: Class lV | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Class at Week 12 and 36
Description: The change from BL in NYHA class at a given visit is a three-category ordinal variable (improved/unchanged/worsened) with the following definition: 1. Improved, if NYHA class decreases at least one level from BL; 2. Unchanged, if NYHA class is unchanged from BL; 3. Worsened, if NYHA class increases at least one level from BL. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Week 12, Week 36
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | Placebo
Number analyzed (Participants) | 9 | 8 | 13 | 18
Participants
  Week 12: Improved | 1 | 1 | 1 | 4
  Week 12: Unchanged | 8 | 7 | 12 | 13
  Week 12: Worsened | 0 | 0 | 0 | 1
  Week 36: number analyzed (Participants) | 3 | 0 | 1 | 3
  Week 36: Improved | 0 | 0 | 0 | 0
  Week 36: Unchanged | 3 | 0 | 1 | 3
  Week 36: Worsened | 0 | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) at Week 36
Description: Evaluation of NT-proBNP was performed by a central laboratory. For Change from baseline, Geometric mean is the geometric mean of the endpoint to baseline ratio. Pre-planned statistical analysis was not performed for this secondary endpoint due to early study termination. Only descriptive statistics are presented.
Time Frame: Baseline, Week 36
Population: The Full Analysis Set (FAS) consisted of all randomized patients who were not mis-randomized. LIK066 doses and placebo arms are considered per study objective. Due to early termination of the study, only the data shown was available.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | Placebo
Number analyzed (Participants) | 3 | 0 | 1 | 3
ratio | 0.7 [0.4 to 1.4] |  | 1.3 [NA to NA] — N/A = there is no upper/lower limit for n = 1 | 1.0 [0.5 to 1.8]

24. Secondary Outcome: Change From Baseline in 24 Hour Urinary Calcium Excretion at Weeks 12 and 36
Description: Urinary calcium excretion was measured from a 24h urine collection from about 25% of randomized patients and analyzed at a central laboratory. Only descriptive analysis done.
Time Frame: Baseline, Week 12, Week 36
Population: Safety Set: All patients who received at least 1 dose of double-blind study drug & included patients who participated in sub-study. Due to early termination of study, only data shown was available. 'Overall Number of Participants Analyzed' = enrolled in 24h urine collection sub-study. 'Number Analyzed '= number of participants with data available
Measure: Mean (Standard Deviation); unit: millimoles per day (mmol/d)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 5
millimoles per day (mmol/d)
  Change from BL at Week 12 | 1.40 (NA) — NA: Not estimable due to insufficient number of participants with events | 3.80 (NA) — NA: Not estimable due to insufficient number of participants with events | 0.10 (0.566) | 0.60 (NA) — NA: Not estimable due to insufficient number of participants with events | -0.49 (3.202)
  Change from BL at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: 24 Hour Urinary Phosphate Excretion at Weeks 12 and 36
Description: Urinary phosphate excretion was measured from a 24h urine collection from about 25% of randomized patients and analyzed at a central laboratory. Only descriptive statistics were done.
Time Frame: Baseline, Week 12, Week 36
Population: The Safety Set (SAF), which consisted of all patients who received at least one dose of double-blind study drug, was considered. The analysis included patients who participated in the 24h urine collection sub-study. Due to early termination of the study, only the data shown was available.
Measure: Mean (Standard Deviation); unit: millimoles per day (mmol/d)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 6
millimoles per day (mmol/d)
  Change from BL at Week 12 | 55.35 (25.809) | 19.25 (55.225) | -125.95 (105.571) | 5.30 (NA) — NA: Not estimable due to insufficient number of participants with events | 26.07 (142.536)
  Change from BL at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) at Weeks 12 and 36
Description: To evaluate bone mineral density as assessed by bone mineral content after 12 weeks and after 36 weeks of treatment. Only descriptive statistics were done.
Time Frame: Baseline, Week 12, Week 36
Population: The Safety Set (SAF), which consisted of all patients who received at least one dose of double-blind study drug, was considered. The analysis included participants who participated in the DXA sub-study. Due to early termination of the study, only the data shown was available.
Measure: Mean (Standard Deviation); unit: grams (g)
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 1
grams (g)
  Wk 12 Whole Body - Hd Hologic Chge BL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Wk 12 Whole Body - Hd Hologic Chge BL | -13.250 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |  | -3.340 (NA) — NA: Not estimable due to insufficient number of participants with events
  Wk 36 Whole Body - Hd Hologic Chge BL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  Wk 36 Whole Body - Hd Hologic Chge BL | -58.220 (NA) — NA: Not estimable due to insufficient number of participants with events |  |  |  | 64.620 (NA) — NA: Not estimable due to insufficient number of participants with events
  Wk 12 Whole Body - Hd Lunar Chge BL: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0
  Wk 12 Whole Body - Hd Lunar Chge BL |  |  | -78.750 (NA) — NA: Not estimable due to insufficient number of participants with events | 37.350 (NA) — NA: Not estimable due to insufficient number of participants with events |
  Wk 36 Whole Body - Hd Lunar Chge BL: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 253 days. Treatment emergent AEs are represented for the double-blind period (i.e., starting from randomization to the end of the double-blind period). Total duration of the double-blind period was planned for approximately 36 weeks.
Arm/Group | LIK066 2.5mg | LIK066 10mg | LIK066 50mg | EMPA 25mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/16 | 0/30 | 0/30 | 1/33
Serious Adverse Events (participants affected / at risk) | 2/15 | 2/16 | 3/30 | 5/30 | 3/33
Other Adverse Events (participants affected / at risk) | 7/15 | 6/16 | 8/30 | 12/30 | 9/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 2.5mg (N=15) | LIK066 10mg (N=16) | LIK066 50mg (N=30) | EMPA 25mg (N=30) | Placebo (N=33)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Cardiac death (General disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Cerebral vascular occlusion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 2.5mg (N=15) | LIK066 10mg (N=16) | LIK066 50mg (N=30) | EMPA 25mg (N=30) | Placebo (N=33)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Genital infection fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 2 | 3 | 1

LIMITATIONS AND CAVEATS:
Due to early discontinuation of the study, the analysis of efficacy was done on the available data (mostly for Epoch 3 (double-blind period 1) only). Because of the small sample sizes the interpretation of the results remained limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT03152552/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03152552/SAP_001.pdf